CLINICAL TRIAL: NCT03833102
Title: Prospective Study of Staphylococcus Aureus Clinical Isolates Versus Colonization: RNAs as Potential Biomarkers for Bloodstream Infections
Acronym: PROSAC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_9726_PROSAC
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — isolates from patients' blood or nostrils
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colonized patients' group (CPG): all adult patients hospitalized in or consulting the Rennes University Hospital, known as S. aureus colonized could be included. In our institution, S. aureus colonization in the nostrils is screened in all patients supposed to undergo neurosurgical or orthopedic surgery.
  Interventions: Other: biological analysis
- SAB patients' group (SAB): all adult patients with SAB could be included. S. aureus colonization in the nostrils will be systematically screened immediately after the first result of positive S. aureus blood culture. Two subgroups will be individualized depending on the SOFA Score:
  * Severe patients
  * Non-severe patients
  Interventions: Other: biological analysis

INTERVENTIONS:
Other: biological analysis — ST types will be determined for all individualized bacterial strains. For all the bacterial strains, RNAs expression will be analyzed at three different growth phases: early exponential phase, mid exponential phase and early stationary phase. Expression of RNAIII and SprD will be evaluated by quantitative polymerase chain reaction.

SUMMARY:
The primary objective is to demonstrate that the risk of S. aureus bacteremia (SAB) is correlated to the RNA III and SprD RNAs expression

DETAILED DESCRIPTION:
Staphylococcus aureus ranks among the top three organisms for community-acquired, healthcare-related and nosocomial infections in humans. It lives as a commensal organism but can also provoke very severe diseases. Identifying markers of the 'colonization/disease' transition is of paramount importance. We recently found that an association of two regulatory RNAs was associated with S. aureus infection rather than colonization and with the severity of infection. Those preliminary results have to be confirmed with a more important prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Patients hospitalized at the University Hospital of Rennes, with according to groups:

  1. : Colonized subjects:

     * Any patient hospitalized at the University Hospital of Rennes, or any health professional, in whom a colonization screening with S. aureus is performed in routine care and a colonization with S. aureus is documented;

     (For information, this screening is carried out frequently at the University Hospital of Rennes for different reasons (before surgery or procedure requiring the installation of equipment, screening of contact cases of infected cases, investigation during a nosocomial epidemic...). These people are hospitalized for reasons other than S. aureus infection and in different departments, but the samples are collected centrally in the institution's bacteriology laboratory.)
  2. : Patients hospitalized for BSA:

     * Patients hospitalized in the infectious diseases and medical intensive care unit and in the surgical intensive care unit, for whom a BSA is documented at the bacteriology laboratory of the University Hospital of Rennes;
     * Patients for whom nasal carrying screening for S. aureus is prescribed as part of their management;
     * These patients will be classified into two groups:

       1. Serious clinic (CG):
* BSA ;
* Associated with signs of sepsis according to the 20168 international definition:

  * SOFA score (see Appendix 3) 2 ;
  * Septic shock will be defined as the existence of sepsis associated with persistent low blood pressure requiring the administration of vasopressors to obtain an average blood pressure (MAP) 65 mmHg and an arterial lactate dosage 2 mmol/L despite adequate vascular filling.

    2) Non-serious clinic (CNG):
* BSA ;
* Which does not meet the definition of the CG group.
* Having expressed their opposition to this research or whose trusted person does not oppose the research if the patient is not able to give an informed opinion.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Persons of full age who are subject to legal protection (protection of justice, guardianship, guardianship), persons deprived of their liberty;
* S. aureus strain producing leucocidin from Panton-Valentine;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized S. aureus colonized or with SAB
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Levels of RNAIII expression and sprD in isolated strains of S. aureus from bacteremia | through study completion, an average of 1 year
  Levels of expression of RNAIII and sprD in isolated strains of S. aureus isolated from bacteremia, compared to these same levels of expression in strains from colonized, uninfected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu REVEST, Principal Investigator — Centre Hospitalier Universitairede Rennes
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France